CLINICAL TRIAL: NCT01891253
Title: Feasibility of the Non-invasive Determination of Cardiac Output Using Inert Gas Rebreathing in Ventilated Patients
Brief Title: Inert Gas Rebreathing in Ventilated Patients
Acronym: VIGR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Joachim Saur, Priv.-Doz. Dr. med., Universitätsmedizin Mannheim
Other Study IDs: VIGR_MA
Record Dates: First submitted 2013-06-20; First posted 2013-07-03 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Sepsis; Respiratory Failure; Heart Failure; Renal Failure
Keywords: cardiac output; mechanical ventilation; inert gas rebreathing; pulse contour analysis
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency; Heart Failure; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ventilated patients: ventilated patients in an internal medicine ICU with existing PiCCO invasive hemodynamic monitoring
  Interventions: Device: non-invasive determination of cardiac output

INTERVENTIONS:
Device: non-invasive determination of cardiac output

SUMMARY:
Measuring hemodynamic parameters in ventilated patients is important yet still complicated to perform. Inert gas rebreathing (IGR) showed promising results when being compared to other invasive as well as non-invasive techniques for the measurement of cardiac output. The aim of our study is to evaluate the feasibility of IGR in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 80 years
* mechanically ventilated patient
* existing PiCCO arterial line

Exclusion Criteria:

* FiO2 > 60% (fraction of inspired oxygen)
* PEEP > 10 mmHg (positive end-expiratory pressure)
* SO2 < 90% (oxygen saturation )
* Systolic blood pressure < 90 mmHg
* Heart rate > 150 bpm
* APRV (airway pressure release ventilation)
* ICD (implantable cardioverter defibrillator) / pace maker
* [ Anaesthetic Conserving Device (Anaconda) ]

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ventilated ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
cardiac output | 1 day
  Determination of cardiac output using invasive pulse contour analysis (PiCCO) and non-invasive inert gas rebreathing (Innocor)

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Saur, MD, Principal Investigator — Universitätsmedizin Mannheim
Locations (1):
- Universitätsmedizin Mannheim, Manheim, Baden-Wurttemberg, Germany